CLINICAL TRIAL: NCT06731803
Title: NeoART - A Phase Ib/II Platform Trial Evaluating the Safety and Activity of Neoadjuvant Trastuzumab-deruxtecan Containing Combination Therapies for HER2+, Resectable Esophagogastric Adenocarcinoma
Brief Title: Platform Trial Evaluating Treatment of Neoadjuvant Trastuzumab-deruxtecan Containing Combination Therapies for HER2+, Resectable Esophagogastric Adenocarcinoma
Acronym: NeoART
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NeoART; 2024-518841-12-00 (EU CTIS Number); AIO-STO-0124 (Other: AIO); IKF072 (Other: IKF Trial ID)
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-12

CONDITIONS: Esophagogastric Adenocarcinoma
Keywords: gastric adenocarcinoma; GEJ adenocarcinoma; Her2 positive
MeSH Terms: interventions — trastuzumab deruxtecan

STUDY DESIGN:
Intervention Model Description: All eligible patients in cohort NeoART-001 will receive: Trastuzumab-deruxtecan 5.4 mg/kg i.v., on day 1, Q3W plus 5-FU/LV: leucovorin 200 mg/m2 i.v., followed by 5-fluorouracil (5-FU) 2600 mg/m2 as a 24-h continuous infusion on day 1, Q2W All eligible patients in cohort NeoART-002 will receive: Trastuzumab-deruxtecan 5.4 mg/kg i.v., on day 1, Q3W plus FLO: oxaliplatin 85 mg/m2 & leucovorin 200 mg/m2, each as an i.v. infusion followed by 5-FU 2600 mg/ m2 as a 24-h continuous infusion on day 1, Q2W followed by surgery determined by the location of the primary tumor and post-operative care according to the guidelines and to local standards outside of this trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NeoART-001 (Experimental): Trastuzumab-deruxtecan 5.4 mg/kg i.v., on day 1, Q3W plus 5-FU/LV: leucovorin 200 mg/m2 i.v., followed by 5-fluorouracil (5-FU) 2600 mg/m2 as a 24-h continuous infusion on day 1, Q2W. Patients will receive three cycles of neoadjuvant T-DXd combined with four cycles 5-FU/LV followed by surgery.
  Interventions: Drug: Trastuzumab deruxtecan + 5FU/LV
- NeoART-002 (Experimental): Trastuzumab-deruxtecan 5.4 mg/kg i.v., on day 1, Q3W plus FLO: oxaliplatin 85 mg/m2 & leucovorin 200 mg/m2, each as an i.v. infusion followed by 5-FU 2600 mg/ m2 as a 24-h continuous infusion on day 1, Q2W. Patients will receive three cycles of neoadjuvant T-DXd combined with four cycles 5-FU/LV followed by surgery.
  Interventions: Drug: Trastuzumab deruxtecan + FLO

INTERVENTIONS:
Drug: Trastuzumab deruxtecan + 5FU/LV — trastuzumab deruxtecan 5.4 mg/kg i.v., on day 1, Q3W for max 3 cycles plus 4 cycles 5-FU/LV: leucovorin 200 mg/m2 i.v., followed by 5-fluorouracil (5-FU) 2600 mg/m2 as a 24-h continuous infusion on day 1, Q2W for 4 cycles
  Arms: NeoART-001
Drug: Trastuzumab deruxtecan + FLO — trastuzumab deruxtecan 5.4 mg/kg i.v., on day 1, Q3W for max 3 cycles plus 4 cycles FLO: oxaliplatin 85 mg/m2 and leucovorin 200 mg/m2, each as an i.v. infusion followed by 5-FU 2600 mg/ m2 as a 24-h continuous infusion on day 1, Q2W for 4 cycles
  Arms: NeoART-002

SUMMARY:
The study is a phase Ib/II, prospective, single arm, open label, non-randomized, multi-center platform trial assessing the feasibility and safety of different neoadjuvant trastuzumab-deruxtecan containing combinational treatment regimens in patients with HER2 positive, locally advanced, resectable esophagogastric adenocarcinoma

DETAILED DESCRIPTION:
The NeoART trial consists of cohorts focusing on distinct trastuzumab-deruxtecan (T-DXd) combination therapies. Enrolment of patients in the two currently defined cohorts will be consecutive, i.e., recruitment for NeoART-002 will start after full recruitment of NeoART-001.

All eligible patients in NeoART-001 cohort will receive: Trastuzumab-deruxtecan 5.4 mg/kg i.v., on day 1, Q3W plus 5-FU/LV: leucovorin 200 mg/m2 i.v., followed by 5-fluorouracil (5-FU) 2600 mg/m2 as a 24-h continuous infusion on day 1, Q2W. Patients will receive three cycles of neoadjuvant T-DXd combined with four cycles 5-FU/LV followed by surgery. Surgery will be scheduled 3-4 weeks after completion of the last cycle of preoperative study therapy.

All eligible patients in NeoART-002 cohort will receive: Trastuzumab-deruxtecan 5.4 mg/kg i.v., on day 1, Q3W plus FLO:oxaliplatin 85 mg/m2 & leucovorin 200 mg/m2, each as an i.v. infusion followed by 5-FU 2600 mg/ m2 as a 24-h continuous infusion on day 1, Q2W. Patients will receive three cycles of neoadjuvant trastuzumab-deruxtecan combined with four cycles FLO followed by surgery.

Surgery will be scheduled 3-4 weeks after completion of the last cycle of preoperative study therapy.

The primary objective of the trial is to evaluate the feasibility and safety (primary endpoint: feasibility rate) of different neoadjuvant T-DXd containing combinational treatment regimens in patients with HER2 positive, locally advanced, resectable esophagogastric adenocarcinoma. The secondary objectives are to futher characterize the efficacy of different neoadjuvant trastuzumab-deruxtecan containing combinational treatment regimens and to evaluate safety and tolerability of different neoadjuvant T-DXd containing combinational treatment regimens. Secondary endpoints comprise the assessment of toxiticy, Perioperative morbidity, Pathological complete remission and R0 resection rate.

Up to 18 patients will be enrolled into each cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Patient* has given written informed consent.
2. Patient is ≥ 18 years of age at time of signing the written informed consent.
3. Patient has histologically proven locally advanced (cT2-4, any cN, M0 OR any cT, cN+, M0 stage) gastric, esophagogastric junction or lower esophageal adenocarcinoma that:

   1. Is considered technically resectable
   2. Does not involve distant site of the peritoneal cavity

      * confirmed by diagnostic laparoscopy for all patients with tumors located in the stomach and those with type 2 and 3 GEJ adenocarcinomas according to guideline recommendation [Lordick et al. 2022].
      * Type 1 GEJ and lower esophageal tumors can be enrolled without diagnostic laparoscopy (which is in line with guidelines and the current routine practice in Germany)
4. Patient has a HER2 positive tumor (by local testing) defined by HER2 IHC 3+ or IHC 2+ plus ISH positive with a HER2:CEP17 ratio of ≥ 2 according to classically used criteria for defining HER2 positivity [Lordick et al. 2017] .
5. Patient has a ECOG performance status 0 or 1.
6. Patient has adequate blood count, liver-enzymes, and renal function:

   1. ANC > 1,500 cells/μL without the use of hematopoietic growth factors
   2. Platelet count ≥ 100 x 109/L (>100,000 per mm3)**
   3. Hemoglobin ≥ 9 g/dL**
   4. Serum total bilirubin ≤ 1.5x institutional upper normal limit (ULN)
   5. AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional ULN
   6. Patients not receiving therapeutic anticoagulation must have an INR ≤ 1.5 ULN and aPTT ≤ 1.5 ULN. The use of full dose anticoagulants is allowed as long as the INR or PTT is within therapeutic limits (according to the medical standard in the institution) and the patient has been on a stable dose for anticoagulants for at least three weeks at the time of inclusion
   7. Serum Creatinine ≤ 1.5 x ULN and a calculated creatinine clearance rate ≥ 50 mL /min
7. Female patients defined as women of childbearing potential (WOCBP) must agree to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of <1% per year during the treatment period and for 6 months after last dose of chemotherapy or 7 months after the last dose of T-DXd, whatever is later.
8. Male patients with WOCBP partners must agree to remain abstinent (refrain from heterosexual intercourse) or use barrier contraceptive during the treatment period as well as up to 4 months after last dose of T-DXd or up to 6 months after last dose of chemotherapy, whatever is later. Male patients must refrain from donating sperm during this same period.

Exclusion Criteria:

1. Patient received previous (radio)chemotherapy or HER2-targeted therapy for the same condition or within the past five years for any other cancerous condition.
2. Patient received prior partial or complete esophagogastric tumor resection.
3. Patient has known hypersensitivity to any component of the T-DXd formulation as well as a known history of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion protein and/or any known contraindication (including hypersensitivity) to one of the study drugs.
4. Patient has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
5. Patient has lung-specific intercurrent clinically significant illnesses including, but not limited to, any underlying pulmonary disorder (e.g., pulmonary emboli within three months of the study enrolment, severe asthma, severe COPD, restrictive lung disease, pleural effusion etc.).
6. Patient received a prior complete pneumonectomy
7. Patient has inadequate cardiac function (LVEF value < 50 %) as determined by echocardiography.
8. Patient has a known complete absence of dihydropyrimidine dehydrogenase (DPD) activity
9. Patient received treatment with brivudine, sorivudine or their chemically related analogues within 28 days prior to stud enrollment
10. Patients has pernicious anemia or other megaloblastic anemia due to vitamin B12 deficiency
11. Patient has peripheral sensitive neuropathy with functional deficits.
12. Patient has a medical history of myocardial infarction (MI) within 6 months before enrollment, symptomatic congestive heart failure (CHF) (New York Heart Association Class II to IV). Subjects with troponin levels above ULN at screening (as defined by the manufacturer), and without any MI related symptoms should have a cardiologic consultation during screening to rule out MI.
13. Patient has a corrected QT interval (QTc) prolongation to > 470 ms (females) or >450 ms (males) based on average of the screening triplicate12-lead ECG.
14. Patient has a history of malignancy other than EGA except for:

    1. Malignancy treated with curative intent and with no known active disease ≥ 5 years before the first dose of study treatment and of low potential risk for recurrence.
    2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
    3. Adequately treated carcinoma in situ without evidence of disease.
15. Patient has an uncontrolled infection requiring IV antibiotics, antivirals or antifungals
16. Patient has active primary immunodeficiency, known uncontrolled active HIV infection or active hepatitis B or C (HBV/HCV) infection. Patients positive for HCV antibody are eligible only if PCR is negative for HCV RNA. Subjects with past or resolved HBV infection are eligible only if they meet all of the following criteria*:

    * HBsAg(-) (for > 6 months off anti-viral treatment)
    * Anti-HBc(+) (IgG or total Ig)
    * HBV DNA undetectable
    * Absence of cirrhosis or fibrosis on prior imaging or biopsy
    * Absence of HCV co-infection or history of HCV co-infection
    * Access to a local hepatitis B expert during and after the study
17. Patient has any autoimmune, connective tissue or inflammatory disorders (e.g., Rheumatoid arthritis, Sjogren's, sarcoidosis etc.) with a documented or suspected pulmonary involvement
18. Patient received live, attenuated vaccine within 30 days prior initiation of study drug
19. Patient has any other serious concomitant or medical condition that, in the opinion of the investigator, presents a high risk of complications to the patient or reduces the likelihood of clinical effect.
20. Patient participated in another interventional clinical study within 28 days prior to study enrollment or participation in a clinical study at the same time as this study, unless it is an observational/ non-interventional study or during the follow-up period of an interventional study.
21. Patient has taken an investigational drug within 28 days prior to initiation of study drug.
22. Female patients, who are pregnant or breast feeding or planning to become pregnant within 7 months after the end of treatment. Female patients of childbearing potential must have a negative serum pregnancy test result within 7 days prior to initiation of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility rate | 9 weeks
  Feasibility rate, defined as proportion of patients receiving the protocol treatment according to the planned schedule before surgery without occurrence of at least one dose-limiting toxicity (DLT)

SECONDARY OUTCOMES:
Safety and toxicity | up to 7.5 months
  Assessment of safety of the treatment as determined by the incidence, type, causality, frequency, timing and severity of adverse events using NCI CTCAE 5.0 and perioperative morbidity (Clavien-Dindo classification) and mortality
Pathological complete remission | up to 10 weeks
  Efficacy will be assessed by the Pathological complete remission (pCR) rate by local assessment corresponding to the ypT0 ypN0 stage category and R0 resection rate

CONTACTS AND LOCATIONS:
Overall Officials: Salah Al-Batran, Prof. Dr., Study Director — Frankfurter Institut für Klinische Krebsforschung IKF GmbH
Locations (11):
- Germany (11):
  - Charite Universitätsmedizin Berlin, Berlin
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Krankenhaus Nordwest GmbH Institut für Klinisch-Onkologische Forschung (IKF), Frankfurt am Main
  - Universitätsmedizin Halle, Universitätsklinikum Halle (Saale), Halle
  - Hämatologisch-Onkologische Praxis Eppendorf (hope), Hamburg
  - Nationales Centrum für Tumorerkrankungen, Heidelberg
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Leipzig, Leipzig
  - Klinikum rechts der Isar München der TU München, München
  - Klinikum Nürnberg, Nuremberg
  - Universitätsklinikum Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No